CLINICAL TRIAL: NCT01817660
Title: Open Versus Endovascular Repair of Popliteal Artery Aneurysm Trial
Acronym: OVERPAR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to unsuccessful trial accrual
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Alik Farber, Associate Professor of Surgery, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OVERPAR Trial
Record Dates: First submitted 2013-03-21; First posted 2013-03-25 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Popliteal Artery Aneurysm
Keywords: popliteal artery aneurysm; endovascular repair; open surgical repair; comparative study
MeSH Terms: conditions — Popliteal Artery Aneurysm | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open Surgery (Active Comparator): In this arm, patients randomized to open surgical repair of popliteal artery aneurysm (OPAR).
  Interventions: Procedure: Open repair of popliteal artery
- Endovascular Surgical repair (EPAR) (Active Comparator): In this arm, patients randomized to endovascular repair of popliteal artery aneurysm (EPAR).
  Interventions: Procedure: Endovascular repair of popliteal artery

INTERVENTIONS:
Procedure: Open repair of popliteal artery
  Other Names: Open repair.
  Arms: Open Surgery
Procedure: Endovascular repair of popliteal artery
  Other Names: Endovascular repair
  Arms: Endovascular Surgical repair (EPAR)

SUMMARY:
Weakness in the wall of a blood vessel located behind the knee (popliteal artery) which leads to a swelling of this blood vessel (aneurysm) is one of the most common types of arterial aneurysms. It is associated with significant risk of blood clot formation, narrowing of blood vessel which can create a serious threat to individual's health. Currently, approved treatment options for this condition include both open surgical and endovascular stent-graft repairs.

In the open repair procedure, the blood vessel behind the knee is tied up or removed and a small artery is created using a vein on the same leg. This is also called a bypass procedure.

In the endovascular repair, using X-rays, doctors places a stent in the blood vessel. Stent is a small device similar to a thin tube. When it is placed in the right location, your doctor can open it. When stent is opened, it supports weakened blood vessel and blood goes through it. The weakened artery then shrinks around the stent.

The OVER-PAR is a short name for this study. Many hospitals in the United States agreed to participate in this study. Patients are randomized to undergo either open or endovascular repair because they can be treated with either of the procedures. Investigators use the short names OPAR for open surgical repair and EPAR for endovascular repair. People who have an aneurysm that is larger than 2 cm (about an inch) can participate in this study.

The purpose of this study is to compare outcomes after these two standard procedures.

DETAILED DESCRIPTION:
Current therapy for patients with asymptomatic PAA, elective repair has been recommended for PAA > 2 cm and for smaller aneurysms with associated mural thrombus1. Treatment modalities are similar in that they exclude the aneurysm from the circulation. Current treatment options include both open surgical bypass (OPAR) with aneurysm exclusion and endovascular popliteal artery repair (EPAR) in which the PAA is excluded by a stent graft. Open repair of PAA has been shown to have excellent graft patency and limb salvage rates, however it is associated with the need for general or regional anesthesia, 10-20% surgical site infection rate, and other complications such as seroma, hematoma, and neurological injury. Endovascular popliteal aneurysm repair is a minimally invasive technique that can be performed under conscious sedation but may be associated with higher risk of graft thrombosis, stent fracture, and may have a lower long term success rate. A paucity of strong comparative data further increases this equipoise. An adequately powered, prospective, comparative study contrasting OPAR approach with EPAR will guide vascular specialists in their treatment of PAA and is very much needed.

Trial Conduct The trial will be conducted in compliance with the protocol, Good Clinical Practice (GCP) guidelines, Declaration of Helsinki and applicable federal regulatory requirements [Title 21 Code of Federal Regulations Parts 50, 54, 56, 812 and 45CFR46]. This trial will be registered on NIH clinical trial registry.

Description and Importance of the Population to be Studied One hundred and forty eights subjects aged 35 or older with asymptomatic ≥ 2.0 cm PAA undergoing repair will be randomized to undergo either OPAR or EPAR. These patients will be recruited at the participating VSGNE centers who agreed to enroll and randomize patients for this trial. This trial will be formally approved by respective Institutional Review Boards.

Investigators will focus on a population of subjects who are candidates for both open surgery and endovascular therapy as determined by the treating investigator. Such individuals represent patients who fall into the "grey area of treatment equipoise". Investigators will exclude subjects with associated acute limb ischemia and hyper-coagulable states. In the OPAR group the choice of conduit will be at the discretion of the surgeon. Vein or non-autogenous conduits will be allowed. In the EPAR group, a femoral cu-down for introduction of stent will be permissible. Percutaneous placement of stent-grafts will also be allowed. Investigators will exclude individuals who are deemed to be at prohibitive risk for open vascular surgery by standard American Heart Association AHA criteria as noted on formal preoperative evaluation or who have significant non-dialysis dependent renal dysfunction (Cr. >3.0). From an anatomic standpoint, investigators will exclude patients who cannot have their PAA treated by stent-grafts due to short "proximal or distal landing zones". Subjects without a patent outflow target vessel will, likewise, be excluded, as treatment options in such patients are usually limited to medical management, amputation or experimental therapies.

TRIAL OBJECTIVES AND PURPOSE

The OVER-PAR Trial is a multicenter randomized trial of best open surgical (OPAR) or best endovascular (EPAR) revascularization in a target population of subjects with asymptomatic ≥ 2.0 cm popliteal artery aneurysm who are candidates for both open and endovascular treatment. The trial has a superiority design and has the following specific aims and hypotheses:

Trial Design The OVER-PAR Trial is a prospective, randomized, open label (two-arm), multicenter, superiority trial comparing the effectiveness of open surgical bypass (OPAR) and endovascular popliteal artery stent graft repair (EPAR) in 148 patients (n=74 in each group) with asymptomatic, clinically significant PAA. Patients with asymptomatic PAA will be screened. These patients will be enrolled from VSGNE centers who agreed to participate in this trial. The proposed trial duration is 4 years. The estimated mean follow-up per subject will be 2.5 years. The trial is powered at 80% to detect a hazard ratio of 1.53, depending on crossover rates, and assuming 2% loss to follow-up.

The Randomization Scheme The randomization scheme will be set up at Boston Medical Center. Participating sites will have access to it by telephone. It is important to emphasize that both procedures to which patients will be randomized are acceptable modalities of care to treat PAA. Within each cohort, subjects will be randomized in a 1:1 ratio to one of the 2 treatment arms by study coordinator at each center. Randomization will follow the following scheme. For each center, sealed, opaque envelopes indicating either OPAR or EPAR repair will be placed in a container in blocks of 6. Each block of 6 envelopes will contain 3 representing OPAR and 3 representing EPAR. When a participating site recruits a patient, a phone call will be made to the central study coordinator at BMC who will open an envelope from the container corresponding to the center and relay the result (OPAR or EPAR) to the coordinator at the requesting center.

Subjects cannot be randomized on the day of surgery since both procedures require some pre-operative planning. For example, a patient who undergoes open repair will need a pre-operative vein mapping to access suitability of vein conduit. Similarly, the patient awaiting EPAR will require procurement of appropriately sized patient-tailored stent -graft for repair of PAA.

Since randomization will be performed during the pre-operative period, the patient will be aware of the surgical plan (open vs. endovascular) prior to the date of the surgery. He or she will then have an option to withdraw from the study and choose any appropriate treatment modality, if they so choose. Additionally, if the surgeon, based on his judgment, decides to offer his patient a different treatment modality from that assigned by the randomization scheme the subject will become a screening failure. Data from subjects categorized as a screening failure will be recorded in the usual registry arm of the VSGNE and used in post-hoc analyses after study completion.

Each subject will be followed for a minimum of 24 months following randomization. Follow-up will continue during the accrual period and therefore the earliest enrolled surviving subject will have a maximum of 48 months follow-up.

Since randomization will be performed during the pre-operative period, the patient will be consulted about the surgical plan (open vs. endovascular) prior to the date of the surgery. He or she will then have an option to withdraw from the study and choose any appropriate treatment modality, if they so choose.

Additionally, if the surgeon, based on his bias, decides to offer his patient a different treatment modality from that assigned by the randomization scheme the subject will become a screening failure.

Subject Withdrawal Criteria

Subjects may be withdrawn from the study for the following reasons:

* Subject declines further study participation.
* In the investigator's judgment, it is in the subject's best interest.

All protocol-specified visits and follow-up procedures should be performed for every subject enrolled in the trial. If the subject refuses to continue with the study visits, every attempt should be made to continue contact by telephone, written communication, or record review to determine if outcome events have occurred, unless the subject specifically refuses such follow-up. The reason for withdrawal will be documented for all subjects withdrawn from the study. If the withdrawing subject is unwilling to have his/her medical records reviewed until the end of the trial period (to document vital status and cause of death), he/she must submit a written refusal.

TREATMENTS TO BE ADMINISTERED Subjects randomized to OVER-PAR endovascular therapy will receive treatment according to established standard of care for exclusion of PAA by commercially available endovascular sten-graft. Subjects receiving endovascular stent-graft(s) will be treated according to the Instructions for Use for the implanted device(s).

Medications/Treatments Permitted and Not Permitted during the Trial There are no medications dispensed specifically for this trial. Investigators should follow standard of care guidelines as well as adhere to Contraindications, Warnings, and Precautions published in the instructions for use of each commercially available endovascular stent.

ASSESSMENT OF EFFICACY Specification of the Efficacy Parameters All-cause mortality will be as reported to occur any time after randomization. Perioperative death is the subset occurring with 30 days of the index procedure.

Amputation above the ankle in the index (treated) leg is a standard definition, as reported in surgical notes.

Re-interventions will be reviewed for the primary endpoint only (new bypass graft, jump/interposition graft revision, thrombectomy/ thrombolysis). All re-interventions (hospitalizations) will be recorded, with length of stay (LOS) discharge diagnoses and (coded) procedures performed for the cost-effectiveness analysis.

Functional Status will be assessed using the SF-12 which is widely used in cardiovascular trials and is available in Spanish, French, for use in North American trials.

Quality of Life will be assessed with using VascuQoL questionnaire7 These are standard, validated instruments, available in Spanish and Canadian French as well as English, for this trial

STATISTICS Analysis of the Primary Endpoints The first phase of analysis will include a description of study variables. This step includes generating summary statistics for study characteristics. Summary statistics will be generated and assessed for the total sample size. The quartiles and median time-to-event outcomes (e.g. MALE-free survival, or MALE-POD) will be estimated using the Kaplan-Meier method and will be reported with two-sided 95% confidence intervals for each intervention arm.

The primary efficacy analysis will be an estimation of the hazard ratio comparing time to MALE and all death rates of subjects receiving OPAR to those receiving EPAR treatment using the nonparametric log-rank test. The hazard ratio and its 95% confidence interval will be estimated in a Cox regression model in which time to MALE+all deaths is the dependent variable and intervention is the independent variable.

The primary analysis will be conducted on an intention-to-treat basis (i.e. based on their randomization status), which includes all subjects randomized, after the last subject has been followed for 1-year or are off study.

Analysis of Secondary Outcomes Other time-to-event outcomes, such as amputation-free survival, described in the secondary aim will be analyzed similarly to the primary analysis.

The above analyses will also be run on the per-protocol population (i.e. based on the actual intervention they received).

ELIGIBILITY:
Inclusion Criteria:

1. Age > 35 years
2. Popliteal artery aneurysm > 2 cm in diameter with or without presence of mural thrombus
3. Candidate for either OPAR or EPAR as judged by the treating investigator.
4. Greater than 2 cm length of normal superficial femoral artery distal to the deep femoral artery takeoff and >2 cm length of normal popliteal artery proximal to the first patent tibial artery.
5. Willing to comply with protocol, attend follow-up appointments, complete all study assessments, and provide written informed consent.

Exclusion Criteria:

1. Popliteal artery thrombosis
2. Popliteal artery aneurysm causing symptomatic thromboembolic disease or compressive symptoms.
3. Superficial femoral artery occlusion or distal tibio-peritoneal occlusion
4. Less than 2 cm length of normal artery to accommodate stent graft seal
5. Life expectancy of less than 2 years.
6. Deemed excessive risk for surgical bypass (defined as prohibitive operative risk by formal pre-procedural cardiac risk assessment undertaken by a cardiologist or internist according to established AHA guideline criteria).
7. A documented hypercoagulable state (defined as a known blood disorder associated with venous or arterial thrombosis).
8. Any infrainguinal revascularization procedure on index leg within 12 weeks prior to treatment initiation.
9. Current immune-suppressive medication, chemotherapy or radiation therapy.
10. Absolute contraindication to iodinated contrast due to prior near-fatal anaphylactoid reaction (laryngospasm, bronchospasm, cardiorespiratory collapse, or equivalent) and which would preclude patient from participation in angiographic procedures.
11. Allergy to stainless steel or nitinol.
12. Pregnancy or lactation.
13. Inability or refusal to provide informed consent.
14. Patients who received an investigational drug for peripheral arterial disease within 4 weeks of screening or who participated in another non-observational clinical trial in the prior 30 days.
15. Prior leg bypass on the ipsilateral limb

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-02; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is major adverse limb events-free survival | Patients are expected to be followed for an average of 2.5 years
  Patients are observed and the two groups are compared for lack of major adverse limb events; above ankle amputation of the index limb or major reintervention-new bypass graft, jump/interposition graft revision, or thrombectomy/ thrombolysis.

SECONDARY OUTCOMES:
Clinical Secondary outcomes: | Average follow-up is expected to be 2.5 years
  Composite of Major adverse limb events (MALE) or perioperative death (POD) (death within 30 days of index procedure); freedom from secondary interventions (major and minor) in index leg; number of interventions (major and minor) per limb salvaged; primary, primary- assisted and secondary patency of the sten-graft or bypass; procedure duration; 30-day freedom from periprocedural Major Adverse Cardiovascular Event (a composite of death, myocardial infarction (MI) and stroke): and perioperative complications.
Functional quality of life | Average patient follow-up is expected to be 2.5 years
  Independent living, ambulatory status, Quality of life (QoL) and functional assessments using VascuQol survey
Resource Utilization | Average follow-up of every patient is expected to be 2.5 years.
  Length of stay and discharge to rehabilitation centers.

CONTACTS AND LOCATIONS:
Overall Officials: Alik Farber, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States